CLINICAL TRIAL: NCT05234801
Title: A Retrospective Data Collection Study of the Internal Fixation and Reconstruction of Bones in the Foot & Ankle Using Various Devices: DARCO Heads; CROSS CHECK 3Di; OrthoLoc 3Di
Brief Title: Retrospective Foot and Ankle Data Collection
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1 849
Record Dates: First submitted 2022-01-20; First posted 2022-02-10 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Lower Limb Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DARCO™ Headed Cannulated Screw: Patients who received a device from the DARCO™ Headed Cannulated Screw family of devices during routine lower limb surgery.
  Interventions: Device: DARCO™ Headed Cannulated Screw
- ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System: Patients who received a device from the ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System family of devices during routine lower limb surgery.
  Interventions: Device: ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System
- ORTHOLOCTM 3Di 2 Foot Reconstruction System: CROSSCHECK™ Module: Patients who received a device from the ORTHOLOCTM 3Di 2 Foot Reconstruction System: CROSSCHECK™ Module family of devices during routine lower limb surgery.
  Interventions: Device: ORTHOLOCTM 3Di 2 Foot Reconstruction System: CROSSCHECK™ Module

INTERVENTIONS:
Device: DARCO™ Headed Cannulated Screw — The DARCO™ Headed Cannulated Screw is a multi-size screw system designed to be used over a guide pin or wire with instrumentation to provide interfragmentary compression and stability for bone fracture/fragment fixation.
  Groups: DARCO™ Headed Cannulated Screw
Device: ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System — A multi-indication foot reconstruction solution providing indication specific implants and instruments designed to address the unique demands of the forefoot and midfoot.
  Groups: ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System
Device: ORTHOLOCTM 3Di 2 Foot Reconstruction System: CROSSCHECK™ Module — A comprehensive fixation system consisting of a wide variety of plate options, created with the purpose of stabilization and fixation of fractures, revision procedures, joint fusion and reconstruction of small bones of the feet.
  Groups: ORTHOLOCTM 3Di 2 Foot Reconstruction System: CROSSCHECK™ Module

SUMMARY:
A retrospective post-market data collection study of the following implant devices :

* DARCO™ Headed Cannulated Screw
* ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System
* ORTHOLOCTM 3Di 2 Foot Reconstruction System: CROSSCHECK™ Module

DETAILED DESCRIPTION:
A retrospective post-market data collection study designed to collect safety and performance Standard of Care data on patients who have undergone routine lower limb surgery that involved one of the following implant devices as per the indication for use:

* DARCO™ Headed Cannulated Screw
* ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System
* ORTHOLOCTM 3Di 2 Foot Reconstruction System: CROSSCHECK™ Module

ELIGIBILITY:
Inclusion Criteria:

Patients 18 years or older at the time of index procedure

• Patients who previously received:

* the Charlotte™ MUC Screw System in accordance with the indications for use: for fixation of bone fractures or for bone reconstruction.
* the CROSSCHECKTM in accordance with the indications for use: Stabilization of fresh fractures, revision procedures, joint fusion and reconstruction of small bones of the feet.
* the ORTHOLOC™ 3Di Recon-Midfoot/Flatfoot System in accordance with the indications for use: Stabilization of fresh fractures, revision procedures, joint fusion and reconstruction of small bones of the feet.
* a DARCO™ Headed Cannulated Screw in accordance with the indications for use: for bone fracture fixation and bone fragment fixation.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective data collection from those who have received the interested devices during lower limb surgery at this single centre.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the performance of the devices concerned. | 1 year.
  Device related intra and post operative adverse events
To demonstrate the safety of the devices concerned. | 3 months
  Device related intra and post operative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bing, FRCS, Study Chair — Robert Jones and Agnes Hunt Orthopaedic Hospital
Locations (1):
- The Robert Jones and Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share the raw retrospective data collected from routine clinical assessments following lower limb surgery.